CLINICAL TRIAL: NCT04627259
Title: Validity And Reliability of the Turkish Version of the Thumb Disability Examination
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Feray Karademir, Research Asssistant, Hacettepe University
Other Study IDs: GO 18/205
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Thumb Osteoarthritis; Thumb Injury; Thumb Fracture; Thumb Laceration
Keywords: thumb; thumb pain; thumb function; questionnaire; examination; validation; cultural adaptation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: patients with thumb pain or functional problems
  Interventions: Other: Thumb Disability Examination

INTERVENTIONS:
Other: Thumb Disability Examination — Turkish Version of Thumb Disability Examination. The Turkish Version of Thumb Disability Examination consists of 20 questions related with thumb pain and functionality.

SUMMARY:
Purpose of the study is the validity and reliability of the Turkish version of The Thumb Disability Examination (TDX) so that it would be used as an assessment tool for Turkish thumb patients.

DETAILED DESCRIPTION:
The hand can be used as a very useful instrument that can perform very complex manipulations that require force and precision. In addition, it is specialized for touch and feeling, and it has a great role in perceiving the environment. The most important part that adds functionality to the hand is the thumb. It contributes more than other fingers during thumb grip activities. However, due to many factors such as inflammatory and neurological causes, orthopedic problems such as tendon and ligament injuries, the thumb joints may be loaded above normal. Mechanical stresses over time cause thumb pain and functional disabilities in daily life activities. Symptoms, muscle strength, normal joint movements, and functional conditions of the patients are objectively evaluated in the clinic by various methods. Patient-based questionnaires, such as The Disabilities of the Arm, Shoulder and Hand (DASH) and Michigan Hand Outcome Questionnaire, can evaluate the independence levels and performances of the patients in daily living activities. However, these questionnaires are used in all upper extremity pathologies, and there is no Turkish scale that evaluates only the function of the thumb, pain and patient satisfaction. During the clinical evaluations of patients with thumb complaints, a scale with a higher sensitivity than the DASH questionnaire, with a validity and reliability study that informs us of their performance and pain from the patients' perspective, is needed. Therefore The Thumb Disability Examination (TDX) was created by selecting the items that are suitable for the thumb from the DASH and Michigan Hand Outcome (MHQ) questionnaires. In this study, cultural adaptation of TDX to Turkish cultural will be done. In this process, the questionnaires will be translated from English to Turkish by two different people. A single Turkish translation will be created from these translations. This Turkish survey will be translated into English by two native speakers of English but who speak Turkish very well, and the English questionnaire will be compared with the original survey. In our study, the Turkish version and reliability (internal consistency, test and retest reliability) of the TDX will be evaluated. Voluntary patients who have been diagnosed in the study and applied to Hacettepe University, Faculty of Physiotherapy and Rehabilitation, Hand Surgery Rehabilitation Unit within the last 6 months will be included. Detailed information about the study to be carried out will be given to the patients face to face and if they accept, the informed consent form will be signed. DASH, SF-36, TDX, Beck Depression and Beck Anxiety, Michigan Hand Outcome Questionnaires, pain, normal joint motion, grip strength assessments will be done to patients twice, 3 days apart.The data obtained as a result of the study will help to identify the problems in patients with thumb pain and to show the effectiveness of the treatments from the patient's perspective. We considered that adding the Turkish adaptation of this questionnaire to the literature by making validity and reliability studies will contribute to clinical evaluations. The data obtained as a result of the study will help to identify the problems in patients with thumb complaints and to show the effectiveness of the treatments from the patient's perspective.

ELIGIBILITY:
Inclusion Criteria:

* able to speak, read, understand and write in Turkish
* having thumb pain
* being over the age of 18

Exclusion Criteria:

* mental disorders
* cognitive limitations
* able not to speak, read, understand and write in Turkish
* out of age 18-80 years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Voluntary patients who applied to Hacettepe University, Faculty of Physiotherapy and Rehabilitation, Hand Surgery and Rehabilitation Unit within the last 6 months, with a history of TMC OA, De Quervain, trigger finger, fracture involving the thumb bones, ligament and tendon injuries, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
Thumb Disability Examination (TDX) | Baseline- 3 days later
  TDX is a 20-question survey divided into 3 sections. It can be calculated as a whole or for each section alone. All scoring is done on a 0-100 scale, with 0 being the least and 100 the most disability.
Visüel Analog Scale- Pain | Baseline
  The severity of the pain felt by individuals during the activity that they have difficulty will be evaluated using the Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline- 3 days later
  DASH contains 30 items related to symptoms and activities of daily living. The total score is 100 and higher scores indicate more disability.

OTHER OUTCOMES:
Michigan Hand Outcomes Questionnaire | Baseline
  It consists of 6 subtitles: general hand function, ADL (unilateral and bilateral), work, pain, aesthetics and satisfaction. Subheadings are filled separately for the right and left hand. The score for each title is calculated separately. The percentage of raw scores obtained by summing the scores given to each question is calculated and normalized. High scores indicate better functional level.
Short Form-36 | Baseline
  Includes 36 questions in eight sub-scales: physical function, physical role restriction, emotional role restriction, body pain, social function, mental health, vitality, and general health. The score of each sub-dimension ranges from 0 to 100. The score is directly proportional to the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Physiotherapy and Rehabilitation Faculty, Hand Surgery Rehabilitation Unit, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Noback PC, Lombardi JM, Seetharaman M, Lee DH, Strauch RJ, Rosenwasser MP. Development and Validation of a Disease-Specific Questionnaire for Basal Joint Arthritis. J Wrist Surg. 2017 May;6(2):126-133. doi: 10.1055/s-0036-1593612. Epub 2016 Oct 14. PMID 28428914
- [Background] Düger T, Yakut E, Öksüz Ç, et al. Kol, Omuz, El Sorunları (Disabilities of the Arm, Shoulder and Hand-DASH) Anketi Türkçe uyarlamasının güvenirliği ve geçerliği. Fizyoter Rehabil. 2006;17:99-107.
- [Background] Oksuz C, Akel BS, Oskay D, Leblebicioglu G, Hayran KM. Cross-cultural adaptation, validation, and reliability process of the Michigan Hand Outcomes Questionnaire in a Turkish population. J Hand Surg Am. 2011 Mar;36(3):486-92. doi: 10.1016/j.jhsa.2010.11.016. Epub 2011 Feb 4. PMID 21295925